CLINICAL TRIAL: NCT01927822
Title: Factors Influencing the Abortion Interval of Second-trimester Termination of Pregnancy Using Misoprostol
Status: Completed | Type: Observational
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief, Department of Obstetrics & Gynecology, Far Eastern Memorial Hospital
Other Study IDs: 102096-F
Record Dates: First submitted 2013-08-18; First posted 2013-08-23 (Estimated); Last update posted 2015-07-07 (Estimated); Status verified 2015-07

CONDITIONS: Labor Induction
Keywords: termination of pregnancy, abortion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pregnancy: Women who underwent termination of pregnancy at second trimester due to a variety of causes

SUMMARY:
This study aims to analyze the factors influencing the abortion interval of second-trimester termination of pregnancy using misoprostol.

DETAILED DESCRIPTION:
Misoprostol is the primary drug of choice for medical termination. It is not only cheap, but also stable at room temperature and easily available worldwide. It is indicated for the treatment of gastritis, but is widely used off-label for a variety of indications in the practice of obstetrics and gynecology, including medication abortion, induction of labor, and the treatment of postpartum hemorrhage. The optimal dosage and route of administration have not been well defined and vary with physicians. The potency of misoprostol's effect varies with dosage, route of administration and dosing interval; both maternal and fetal factors may, to certain extent, affect the abortion interval. This study aims to analyze the factors influencing the abortion interval of second-trimester termination of pregnancy using misoprostol.

ELIGIBILITY:
Inclusion Criteria:

1.All female patients who were admitted for medical termination of second-trimester pregnancy

Exclusion Criteria:

1. Patients who are allergy to Cytotec.

Ages: 13 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: This is a single-center, retrospective chart review study. All female patients who were admitted for medical termination of second-trimester pregnancy from January 2008 to May 2013, at the Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital were recruited.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2013-08; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Successful termination rate by Cytotec. | 1 week

SECONDARY OUTCOMES:
Factors affecting abortion interval by cytotec. | 1 week
  To identify the factors affecting termination interval Cox regression model.

CONTACTS AND LOCATIONS:
Overall Officials: Sheng-Mou Hsiao, MD, Principal Investigator — Far Eastern Memorial Hospital
Locations (1):
- Far Eastern Memorial Hospital, New Taipei, Taiwan, Taiwan